CLINICAL TRIAL: NCT04137445
Title: The Effects of Early Complementary Feeding on Growth, Neurodevelopment, Sleep and Gut Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-0546; R01DK126710 (NIH)
Record Dates: First submitted 2019-10-17; First posted 2019-10-24 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Linear Growth; Neurodevelopment; Gut Microbiome
Keywords: Complementary Feeding
MeSH Terms: interventions — Infant Food

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Provided Diet (Experimental): A group of complementary foods provided to participants by researchers.
  Interventions: Other: Baby Foods
- Traditional Diet (Placebo Comparator): No study foods provided to participants by researchers. Participants will eat a typical diet provided by caregivers.
  Interventions: Other: Foods from the home

INTERVENTIONS:
Other: Baby Foods — Commercially available baby foods
  Arms: Study Provided Diet
Other: Foods from the home — Caregiver will provide participant with usual foods from the home
  Arms: Traditional Diet

SUMMARY:
The overall objective of this project is to understand how consuming a prescribed diet of different infant foods (which may contain cereals,fruits, vegetables, meats, dairy) during the time of early complementary feeding (~5 to 12 months) in breastfed infants has on growth trajectories, neurodevelopment and sleep patterns in relation to gut microbiota, compared with a traditional diet that is usually provided in the home to infants.

The three primary aims include:

Aim 1: Identify the effects that the prescribed early complementary feeding specific study diet has on growth trajectories in breastfed infants.

Aim 2: Identify whether the relationship between the prescribed early complementary feeding specific study diet and growth is mediated by gut microbiota.

Aim 3: Characterize infant neurodevelopment and sleep patterns.

DETAILED DESCRIPTION:
Some details are intentionally left to out to preserve the scientific integrity of the study, and they will be included in the record after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Full term: gestational age > 37 weeks
* Exclusively breastfed (< 2 weeks of cumulative formula exposure). Any formula consumption on a given day is considered one day of formula exposure. During the intervention, if the participant receives more than 50% of the liquid diet from infant formula, s/he will be excluded from the study.
* Maternal conditions such as gestational diabetes mellitus, preeclampsia, multiple pregnancies are acceptable.

Exclusion Criteria:

* Large for gestational age or small for gestational age
* Antibiotic use from birth to the time of enrollment
* Documented food allergies
* Previous complementary food exposure
* Conditions that would affect protein metabolism or growth

Ages: 5 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Weight | Over 6 months
  Measured in kg
Length | Over 6 months
  Measured in cm
Gut Microbiome | Over 6 months
  Gut microbiota structure by 16S sequencing

SECONDARY OUTCOMES:
Neurodevelopment | At 12 months of age
  Fine motor skills and cognition measured by the Bayley - III
Duration of sleep | Over 6 months
  Measured in minutes per 24 hours by the MicroMini-Motionlogger actigraph
Body composition | Over 6 months
  Body fat mass, fat-free mass measured by stable isotopes
Serum c-reactive protein (CRP-hs) | Over 6 months
  Measured in mg/L
Serum IGF-1 (Insulin-like growth factor1/ somatomedin C) | Over 6 months
  Measured in ng/mL
Serum IGFBP-3 (Insulin-like growth factor-binding protein 3) | Over 6 months
  Measured in ng/mL
Dietary intake | Over 6 months
  3 day dietary recall with results generated by NDSR software
Total calories in breast milk | Over 6 months
  Measured in kcal/100 mL
Total carbohydrates in breast milk | Over 6 months
  Measured in g/100 mL
Total protein in breast milk | Over 6 months
  Measured in g/100 mL
Total fat in breast milk | Over 6 months
  Measured in g/100 mL

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Tang, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Odiase E, Frank DN, Young BE, Robertson CE, Kofonow JM, Davis KN, Berman LM, Krebs NF, Tang M. The Gut Microbiota Differ in Exclusively Breastfed and Formula-Fed United States Infants and are Associated with Growth Status. J Nutr. 2023 Sep;153(9):2612-2621. doi: 10.1016/j.tjnut.2023.07.009. Epub 2023 Jul 26. PMID 37506974